CLINICAL TRIAL: NCT00545558
Title: Antiretroviral Therapy and the Hepatitis C Virus
Brief Title: Effects of Anti-HIV Drugs on the Hepatitis C Virus (HCV) in Adults Infected With Both HCV and HIV
Acronym: ART and HCV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kenneth Sherman, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01AI065256-01 (NIH); 5R01AI065256 (NIH)
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Hepatitis C; HIV Infections
Keywords: Antiretroviral Therapy, Highly Active; Coinfection; Treatment Naive
MeSH Terms: conditions — Hepatitis C; HIV Infections; Coinfection | interventions — efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will receive ART consisting of efavirenz and the co-formulation of emtricitabine and tenofovir disoproxil fumarate. If participants are unable to tolerate the treatment, a different regimen will be prescribed.
  Interventions: Drug: Efavirenz; Drug: Emtricitabine/Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Efavirenz — 600 mg tablet taken orally daily
Drug: Emtricitabine/Tenofovir disoproxil fumarate — 200 mg emtricitabine/ 300 mg tenofovir disoproxil fumarate tablet taken orally daily

SUMMARY:
The purpose of this study is to measure the effects of anti-HIV drugs on hepatitis C virus (HCV) viral load in people infected with both HCV and HIV.

DETAILED DESCRIPTION:
Coinfection with HCV and HIV occurs in 20% to 30% of HIV infected people in the United States. Individuals with HCV/HIV coinfection tend to have higher HCV viral loads than individuals with HCV alone. However, current evidence suggests that initiation of effective antiretroviral therapy (ART) may be associated with increases in HCV viral load. The purpose of this study is to evaluate changes in HCV viral load associated with the initiation of ART in HCV/HIV coinfected adults.

All participants will receive ART consisting of efavirenz once daily and the co-formulation of emtricitabine and tenofovir disoproxil fumarate (DF) once daily. If participants are unable to tolerate a different regimen would be prescribed.

There will be at least 21 study visits. During the first week of the study, participants will undergo blood draws for viral kinetic sampling and initiation of study medications. Following the first week, there will be weekly visits for 96 weeks. At screening, participants will undergo vital signs measurements, a physical exam, medical history, blood collection, and liver biopsy. During Week 1, participants will be hospitalized for 24 hours for initiation of ART and viral kinetic sampling. Blood draws for viral kinetic sampling of HCV and HIV will be performed at Hours 0, 2, 4, 6, 9, 12, 18, and 24. Participants will return to the clinic or hospital at Hours 48, 72, 96, and 167 for additional viral kinetic sampling. Blood collection will occur at all visits; physical exams, vital signs measurement, a side effects questionnaire, and urine and semen collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HCV-infected
* HIV-infected
* Liver biopsy consistent with chronic hepatitis within 1 year of study entry.
* ART-naive or no ART for at least 3 months prior to study entry

Exclusion Criteria:

* Hemoglobin less than 9 g/dl.
* Hepatitis B virus infected or antibody to hepatitis B core antigen, alpha-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, autoimmune disorder, or other concurrent liver disease
* Decompensated liver disease evidenced by active or history of encephalopathy, ascites, or variceal bleeding; prothrombin time (PT) greater than 3 seconds above normal or international normalized ratio (INR) greater than 1.3 sec; platelet count less than 90,000 K/ul. Participants with cirrhosis will not be excluded.
* Active thyroid disease. Participants on thyroid replacement therapy with normal thyroid-stimulating hormone are not excluded.
* Chronic kidney insufficiency, defined as creatinine clearance of greater than approximately 50 ml/min
* Life-threatening disease processes other than HIV or HCV that could interfere with participation in the study
* Any condition that, in the opinion of the investigator, may interfere with completion of the study regimen. This includes severe psychiatric disorders, or active alcohol or recreational drug abuse
* Use of systemic corticosteroids or immunomodulatory drugs within 1 month prior to study entry
* Current or prior successful interferon treatment
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Underlying patterns of liver injury and hepatitis C virus (HCV) viral changes after antiretroviral therapy (ART) initiation | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E. Sherman, MD, PhD, Principal Investigator — Unviersity of Cincinnati
Locations (2):
- United States (2):
  - General Clinical Research Center (GCRC), OH site, Cincinnati, Ohio
  - Virginia Commonwealth University, School of Medicine, Richmond, Virginia

REFERENCES:
- [Background] Shudo E, Ribeiro RM, Perelson AS. Modelling hepatitis C virus kinetics during treatment with pegylated interferon alpha-2b: errors in the estimation of viral kinetic parameters. J Viral Hepat. 2008 May;15(5):357-62. doi: 10.1111/j.1365-2893.2007.00954.x. PMID 18380660
- [Background] Shudo E, Ribeiro RM, Perelson AS. Modelling the kinetics of hepatitis C virus RNA decline over 4 weeks of treatment with pegylated interferon alpha-2b. J Viral Hepat. 2008 May;15(5):379-82. doi: 10.1111/j.1365-2893.2008.00977.x. Epub 2008 Feb 11. PMID 18266841
- [Background] Blackard JT, Sherman KE. HCV/ HIV co-infection: time to re-evaluate the role of HIV in the liver? J Viral Hepat. 2008 May;15(5):323-30. doi: 10.1111/j.1365-2893.2008.00970.x. Epub 2008 Jan 17. PMID 18208497
- [Background] Ma G, Barrett A, Sherman KE, Shata T, Blackard J. Detection of HIV in Liver Biopsies and Intrahepatic Lymphocytes. 15th Conference on Retroviruses and Opportunistic Infections. Boston, MA February 2008
- [Background] Sherman KE, Rouster S, Feinberg J, Bini E, Blackard J, Shata T. Hepatic Apoptosis following Initiation of ART in HCV/HIV co-infected Subjects. 16th Conference on Retroviruses and Opportunistic Infections, Montreal, Canada February 2009
- [Background] Blackard J, Ma G, Rouster S, Martin C, Shata T, Sherman K. Baseline hepatitis C virus variability does not predict flares in HIV/HCV co-infected persons initiating antiretroviral therapy. 5th International Workshop on HIV and Hepatitis Co-infection, Lisbon, Portugal, June 2009.
- [Background] Blackard J, Ma G, Rouster S, Barrett A, Shata T, Sherman K. HIV is frequently detected in liver biopsy tissue. 5th International Workshop on HIV and Hepatitis Co-infection, Lisbon, Portugal, June 2009.
- [Background] Shata MT, Bartholomew KA, Rouster SD, Blackard JT, Sterling RK, Bini E, Perelson AS, Goodman ZD and Sherman KE. Strong HCV and HIV immune responses in coinfected subjects who experienced ALT flare and/or rebound HCV viral load after ART initiation. 17th Conference on Retroviruses and Opportunistic Infections, San Francisco, CA, February 2010.
- [Background] Blackard JT, Ma G, Martin CM, Rouster SD, Shata MT, Sherman KE. HIV variability in the liver and evidence of possible compartmentalization. AIDS Res Hum Retroviruses. 2011 Oct;27(10):1117-26. doi: 10.1089/aid.2010.0329. Epub 2011 May 4. PMID 21417757
- [Result] Sherman KE, Guedj J, Shata MT, Blackard JT, Rouster SD, Castro M, Feinberg J, Sterling RK, Goodman Z, Aronow BJ, Perelson AS. Modulation of HCV replication after combination antiretroviral therapy in HCV/HIV co-infected patients. Sci Transl Med. 2014 Jul 23;6(246):246ra98. doi: 10.1126/scitranslmed.3008195. PMID 25101888